CLINICAL TRIAL: NCT06569836
Title: Evaluation Study for the "Jockey Club E-Generation: Impact Extension Project for Chronic Knee Pain Management"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Sheng Kung Hui Welfare Council Limited (Other)
Responsible Party: Principal Investigator, Dr. Pui-Hing Chau, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AR230018
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Knee Discomfort; Knee Pain Chronic
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned intervention (Other): The intervention group will start the 12-week intervention immediately
  Interventions: Other: 12-week intervention
- Assigned waitlist control (Other): The waitlist control group will have weekly educational and virtual workshops for 12 weeks.
  After 12 weeks assessment, the control group will receive the same intervention as the intervention group for 12 weeks.
  Interventions: Other: 12-week intervention; Other: 12-week attention control

INTERVENTIONS:
Other: 12-week intervention — Rehabilitation Exercise Plan Week 1-4 For No Symptom Group: Therapeutic home exercise prescription(2 sessions, 60 minutes per session) For Mild & Moderate Group: Rehabilitation Plan provided by Physiotherapist (4 sessions, 60 minutes per session)
  Enhancement of Self-Management Capacity Week 5-8 For No Symptom Group: Educational Workshops provided by Physiotherapist (2 sessions, 60 minutes per session) For Mild & Moderate Group: Self-management group provided by Social Worker (4 sessions, 60 minutes per session)
  Exercise Maintenance Week 9-12 For No Symptom Group: Mobilized Intervention (2 sessions, 60 minutes per session) For Mild & Moderate Group: Exercise Maintenance provided by Exercise Mentor (4 sessions, 60 minutes per session)
Other: 12-week attention control — The attention and waitlist control group will have weekly educational and virtual workshops for 12 weeks. Three topics will be covered, including online exercise class, cognitive training, leisure and recreational activities. Each session will be 30-45 minutes and each topic last for four weeks. Participants could access the virtual sessions by their electronic devices.
  Arms: Assigned waitlist control

SUMMARY:
Objectives:

This study aims to evaluate the effectiveness of the "Jockey Club E-Generation: Impact Extension Project for Chronic Knee Pain Management", with a view to developing sustainable strategies of self-management on chronic conditions integrating with tele-rehabilitation technology.

Study design and participants:

An evaluation study adopting a randomized controlled trial design, with waitlist attention control will be conducted in Elderly community centres of Hong Kong Sheng Kung Hui Welfare Council and Christian Family Service Centre (CFSC) in Hong Kong. The proposed sample size is 858 participants, which is a convenience sample from the service user of the "Jockey Club E-Generation: Impact Extension Project for Chronic Knee Pain Management". At least 15 participants will be invited for qualitative interview.

Participants will be randomized to the intervention group or the waitlist attention control group in 1:1 ratio using block randomization with random block size of 4, 6 and 8, stratified by each centre and severity of condition. A researcher independent to the project will generate the randomization sequence by computer and keep the list. Participants in the intervention group (known as Group A to the participants) will start the 12-week intervention immediately, whereas the waitlist attention control (know as Group B to the participants) will start the intervention after 12 weeks. During the waiting period, waitlist control receives attention control.

Measurements:

The primary outcome of this study is quality of life. It will be measured by the Hong Kong Chinese version of World Health Organization Quality-of-Life Scale (WHOQOL-BREF).

The secondary outcomes are pain, physical functioning, emotional functioning, adherence rate, satisfaction score, rate of adverse events in relation to the intervention, and cost-effectiveness of the intervention.

Expected results:

The improvement in health-related quality of life of older adults is larger in the intervention group as compared to the control group; The relief in knee pain of older adults is larger in the intervention group as compared to the control group; The improvement in physical functioning of older adults is larger in the intervention group as compared to the control group; The improvement in emotional functioning of older adults is larger in the intervention group as compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

i. Aged ≥55 years;

ii. Community-dwelling;

iii. With self-reported knee pain problem currently or in the past 12 months;

iv. Cognitively sound (screened by the Clock Drawing Test (CDT) ≤ 4 (Agrell & Dehlin, 1998));

v. Able to understand and communicate in Cantonese or Mandarin.

Exclusion Criteria:

i. Diagnosed with stroke, myocardial infarction, injury or inflammation of the knee, autoimmune disease, unable to walk in the past three months;

ii. Users/ of Hospital Authority medical consultation or physiotherapy or occupational therapy services related to osteoarthritis knee;

iii. Screened to have three or above conditions including significant knee symptom score 5 or above, WOMAC Score ≥48, 5 times Sit to Stand test >16.7 seconds, Time Up and Go Test >14 seconds, Age >80 and BMI >25.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 858 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline quality of life at 12 weeks. | 12 weeks after baseline.
  Measured by the Hong Kong Chinese version of World Health Organization Quality-of-Life Scale (WHOQOL-BREF). Scoring based on a rule set by the World Health Organization and converted to a score between 4 and 20 for all domains, with the higher the score, the better the quality of life.

SECONDARY OUTCOMES:
Change from baseline quality of life at 24 weeks. | 24 weeks after baseline, only for waitlist control group.
  Measured by the Hong Kong Chinese version of World Health Organization Quality-of-Life Scale (WHOQOL-BREF). Scoring based on a rule set by the World Health Organization and converted to a score between 4 and 20 for all domains, with the higher the score, the better the quality of life.
Change from baseline pain at 12 weeks. | 12 weeks after baseline.
  Measured by the pain subscale of Chinese version of Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). Total score ranges from 0 to 96. Higher scores indicate worse pain, stiffness, and functional limitations.
Change from baseline pain at 24 weeks. | 24 weeks after baseline, only for waitlist control group.
  Measured by the pain subscale of Chinese version of Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). Total score ranges from 0 to 96. Higher scores indicate worse pain, stiffness, and functional limitations.
Change from baseline physical functioning, Five Times Sit-to-Stand Test at 12 weeks. | 12 weeks after baseline.
  Measured by the Five Times Sit-to-Stand Test, scoring the amount of time a patient is able to transfer from a seated to a standing position and back to sitting five times. The lower the time to complete the test the better the outcome of the test.
Change from baseline physical functioning, Five Times Sit-to-Stand Test at 24 weeks. | 24 weeks after baseline, only for waitlist control group.
  Measured by the Five Times Sit-to-Stand Test, scoring the amount of time a patient is able to transfer from a seated to a standing position and back to sitting five times. The lower the time to complete the test the better the outcome of the test.
Change from baseline physical functioning, 2-minute Step Test at 12 weeks. | 12 weeks after baseline.
  Measured by the 2-minute Step Test, scoring how many times the patient's right knee reaches the point that is halfway between the midpoint of the patient's patella and the top of their iliac crest while marching in place for 2 minutes. Higher scores indicate greater levels of aerobic capacity.
Change from baseline physical functioning, 2-minute Step Test at 24 weeks. | 24 weeks after baseline, only for waitlist control group.
  Measured by the 2-minute Step Test, scoring how many times the patient's right knee reaches the point that is halfway between the midpoint of the patient's patella and the top of their iliac crest while marching in place for 2 minutes. Higher scores indicate greater levels of aerobic capacity.
Change from baseline emotional functioning, Self-Efficacy to Manage Chronic Disease at 12 weeks. | 12 weeks after baseline.
  Measured by the Self-Efficacy to Manage Chronic Disease Scale, scoring range from 1 to 10, the higher the score, the greater the self-efficacy.
Change from baseline emotional functioning, Self-Efficacy to Manage Chronic Disease at 24 weeks. | 24 weeks after baseline, only for waitlist control group.
  Measured by the Self-Efficacy to Manage Chronic Disease Scale, scoring range from 1 to 10, the higher the score, the greater the self-efficacy.
Change from baseline emotional functioning, Cognitive Symptom Management at 12 weeks. | 12 weeks after baseline.
  Measured by the Cognitive Symptom Management (CSM) Scale, scoring range from 0 to 5, with a higher score indicating more practice of these techniques.
Change from baseline emotional functioning, Cognitive Symptom Management at 24 weeks. | 24 weeks after baseline, only for waitlist control group.
  Measured by the Cognitive Symptom Management (CSM) Scale, scoring range from 0 to 5, with a higher score indicating more practice of these techniques.
Change from baseline emotional functioning, Sleep Quality at 12 weeks. | 12 weeks after baseline.
  Measured by the Pittsburgh Sleep Quality Index (PSQI), scoring range from 0 to 21 with higher score indicating poorer quality.
Change from baseline emotional functioning, Sleep Quality at 24 weeks. | 24 weeks after baseline, only for waitlist control group.
  Measured by the Pittsburgh Sleep Quality Index (PSQI), scoring range from 0 to 21 with higher score indicating poorer quality.
Change from baseline emotional functioning, depression at 12 weeks. | 12 weeks after baseline.
  Measured by the Patient Health Questionnaire-9 (PHQ-9), scoring range from 0 to 27, the higher the score, the more severe the depression.
Change from baseline emotional functioning, depression at 24 weeks. | 24 weeks after baseline, only for waitlist control group.
  Measured by the Patient Health Questionnaire-9 (PHQ-9), scoring range from 0 to 27, the higher the score, the more severe the depression.
Change from baseline emotional functioning, quality of life at 12 weeks. | 12 weeks after baseline.
  Measured by the World Health Organization Quality-of-Life Scale (WHOQOL-BREF), scoring based on a rule set by the World Health Organization and converted to a score between 4 and 20 for all domains, with the higher the score, the better the quality of life.
Change from baseline emotional functioning, quality of life at 24 weeks. | 24 weeks after baseline, only for waitlist control group.
  Measured by the World Health Organization Quality-of-Life Scale (WHOQOL-BREF), scoring based on a rule set by the World Health Organization and converted to a score between 4 and 20 for all domains, with the higher the score, the better the quality of life.
Adherence rate | During 12 weeks intervention
  Collected by a practice record in the App, as well as class attendance record for face-to-face classes
Satisfaction score | 12 weeks after baseline for intervention group, 24 weeks after baseline for waitlist control group.
  Assessed by a five-point Likert scale, 0 indicates not satisfied at all, 4 indicates very satisfied. The higher the score, the higher the satisfaction level.
Rate of adverse events in relation to the intervention | 12 weeks after baseline for intervention group, 24 weeks after baseline for waitlist control group.
  Symptoms and adverse events will be recorded by a single question.
Cost-effectiveness of the intervention | 12 weeks after baseline for intervention group, 24 weeks after baseline for waitlist control group.
  Expenses related to (emergency department visits, outpatient, inpatient, rehabilitation, over-the-counter medication and supplement) related to knee pain or falls will be collected. Costing of the intervention from the service provider will be obtained from the service provider directly.

CONTACTS AND LOCATIONS:
Overall Officials: Pui Hing Chau, PhD, Principal Investigator — School of Nursing, The University of Hong Kong
Locations (1):
- Elderly community centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No